CLINICAL TRIAL: NCT04835415
Title: Ultrasound Guided : Retrolaminar Block Versus Thoracic Epidural Analgesia for Pain Control Following Laparoscopic Cholecystectomy
Brief Title: Ultrasound Guided : Retrolaminar Block Versus Thoracic Epidural Analgesia Following Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Dina Abdelhameed Elsadek Salem, Principle investigator, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6777
Record Dates: First submitted 2021-04-04; First posted 2021-04-08 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Analgesia
Keywords: Ultrasound; Bilateral retrolaminar; Thoracic epidural; post operative analgesia; Laparoscopic cholecystectomy
MeSH Terms: conditions — Agnosia | interventions — Tea

STUDY DESIGN:
Intervention Model Description: Analgesia for postoperative pain after laparoscopic cholecystectomy by using ultrasound-guided retrolaminar block vs ultrasound-guided thoracic epidural analgesia.
Who Masked: Participant, Outcomes Assessor
Masking Description: Double (participant, outcomes assessor) Anesthetist not sharing in the study will assess patient.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group T (Active Comparator): Group (T) (n=26): will receive ultrasound guided thoracic epidural analgesia: 20 ml of bupivacaine 0.25 % plus 5ug/ml adrenaline (1:200000).
  Interventions: Procedure: Thoracic epidural analgesia
- group R (Active Comparator): Group (R) (n=26): will receive bilateral ultrasound guided retrolaminar block analgesia: 20 ml of bupivacaine 0.25 % plus 5ug/ml adrenaline (1:200000).
  Interventions: Procedure: Bilateral retrolaminar block

INTERVENTIONS:
Procedure: Bilateral retrolaminar block — in lateral position and after skin sterilization. The spine is palpated from cervical (C7) downward toT7 and point marked to identify the spinous process. The linear high frequency transducer (6-13 MHz) will be placed parasagittal plane 1 cm lateral to the midline. The needle (18 gauge) is inserted in the plane view of the ultrasound probe to target the T7 and needle is advanced from downward to upward until the needle tip contacted the lamina. After negative aspiration, a 20 ml of bupivacaine 0.25 % plus 5ug/ml adrenaline (1:200000) will be injected. The procedure will be repeated following the same steps on the other side.
  Other Names: Ultrasound guided retrolaminar block
  Arms: group R
Procedure: Thoracic epidural analgesia — In the lateral position, after skin sterilization, Ultrasound with high frequency linear probe (5-13 MHz). Thoracic intervertebral space (T7-8) will be identified by counting from the C7 to prominent thoracic spine (T7). The probe will be used in parasagittal plane 2 cm from midline. The probe will be directed medially to identify the dura matter at the T7-8 intervertebral space . the needle 18 gauage will be inserted in plane to target T7-8 intervertebral space ., after needle tip reached target space, loss of resistance technique then 20 ml bupivacaine 0.25% plus 5ug/ml adrenaline (1:200000) was injected after aspiration
  Other Names: Ultrasound guided thoracic epidural
  Arms: group T

SUMMARY:
The aim of this study is to evaluate analgesic effect of ultrasound-guided retrolaminar block vs ultrasound-guided thoracic epidural analgesia in pain control following laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
To study the difference between the effects of ultrasound-guided bilateral retrolaminar block and ultrasound-guided thoracic epidural analgesia on pain control following laparoscopic cholecystectomy. To relief pain and improve satisfaction in patients undergoing laparoscopic cholecystectomy at Zagazig university hospitals.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent from the patient.
* Age: 21-45 years old.
* Sex: both sex (males and females).
* Physical status: ASA 1& II.
* BMI = (25-35 kg/m2).
* Type of operation: elective laparoscopic cholecystectomy

Exclusion Criteria:

* Altered mental state.
* Patients with known history of allergy to study drugs.
* Advanced hepatic, renal, cardiovascular, and respiratory diseases.
* Patients with chronic pain.
* Patients receiving anticoagulants.
* Contraindications of regional anesthesia, e.g., allergy to local anesthetics, coagulopathy, or septic focus at site of injection.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2021-04-10 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Pain intensity at rest and at cough using Numerical Rating Scales (NRS) | 30 minutes postoperative
  measured by NRS consisted of a series of numbers represents range of pain intensity (10 means the worst pain and 0 means no pain)
Pain intensity at rest and at cough using Numerical Rating Scales (NRS) | at 1 hour postoperative
  measured by NRS consisted of a series of numbers represents range of pain intensity (10 means the worst pain and 0 means no pain)
Pain intensity at rest and at cough using Numerical Rating Scales (NRS) | at 2 hours postoperative
  measured by NRS consisted of a series of numbers represents range of pain intensity (10 means the worst pain and 0 means no pain)
Pain intensity at rest and at cough using Numerical Rating Scales (NRS) | at 4 hours postoperative
  measured by NRS consisted of a series of numbers represents range of pain intensity (10 means the worst pain and 0 means no pain)
Pain intensity at rest and at cough using Numerical Rating Scales (NRS) | at 6 hours postoperative
  measured by NRS consisted of a series of numbers represents range of pain intensity (10 means the worst pain and 0 means no pain)
Pain intensity at rest and at cough using Numerical Rating Scales (NRS) | at 8 hours postoperative
  measured by NRS consisted of a series of numbers represents range of pain intensity (10 means the worst pain and 0 means no pain)
Pain intensity at rest and at cough using Numerical Rating Scales (NRS) | at 10 hours postoperative
  measured by NRS consisted of a series of numbers represents range of pain intensity (10 means the worst pain and 0 means no pain)
Pain intensity at rest and at cough using Numerical Rating Scales (NRS) | at 12 hours postoperative
  measured by NRS consisted of a series of numbers represents range of pain intensity (10 means the worst pain and 0 means no pain)

SECONDARY OUTCOMES:
Time to first call of rescue analgesia | within 12 hours postoperative
  start from retrolaminar or epidural injection of the drug to the time of first call of naluphine
Total analgesic (Naluphine) consumption | within 12 hours postoperative
  Total consumption of rescue analgesia(Naluphine) post operative
The number of participant with complications of the techinque (dural puncture , nerve injury, spinal injection, epidural haematoma, pleural puncture) | within 24 hours postoperative
  The numer of participant with complications of the techinque (dural puncture , nerve injury, spinal injection, epidural haematoma, pleural puncture)
Patient satisfaction is recorded at the end of 24 hours postoperative | 24 hours postoperative
  using 5-point Likert-like verbal rating scale by asking the patient about "how he/she evaluated their experience with the analgesic management after the surgery?"5=very satisfied, 4=satisfied, 3= neutral, 2= dissatisfied and 1= very dissatisfied".
The number of participant with nausea, vomiting, hypotension and bradycardia. | 24 hours postoperative
  the number of participant with nausea (sensation of being about to vomit), vomiting (the expelling of the food content from the stomach through mouth, it will be treated by 4 mg ondansetron), hypotension (if MAP decreases more than 20% of basal reading it will be treated by 12 mg ephedrine) and bradycardia (if HR less than 50 beats/min it will be treated by 0.5 mg atropine).

CONTACTS AND LOCATIONS:
Overall Officials: Dina Salem, MD., Principal Investigator — faculty of medicine , Zagazig University
Locations (1):
- faculty of medicine, Zagazig university, Zagazig, Egypt

IPD SHARING:
Plan to Share IPD: No